CLINICAL TRIAL: NCT00612495
Title: Parallel Randomised Open Phase II Study of Oxaliplatin (L-OHP) Alone and in Combination With 5-Fluorouracil (5-FU) in Patients With Locally Advanced or Metastatic Endometrial Cancer Previously Treated With Cisplatin or Arboplatin
Brief Title: Endometrial Cancer - LOHP Alone and With 5FU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Nathalie Billon/Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC_7496
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Oxaliplatin; Fluorouracil

INTERVENTIONS:
Drug: oxaliplatin, 5 FU — Oxaliplatin:130 mg/m² as a 2-hour intravenous (IV) infusion in 500 mL of 5% glucose solution on Day 1 and repeated every 3 weeks.
  5-FU: following oxaliplatin administration, 1000 mg/m²/day as a continuous IV infusion from Day 1 to Day 4, repeated every 3 weeks.
  Other Names: Eloxatin, Fluorouracil

SUMMARY:
To determine the efficacy (response rate [RR], time to progression and survival) of oxaliplatin as a single agent and oxaliplatin in combination with 5 FU in patients with advanced/metastatic endometrial cancer pretreated with one prior chemotherapy regimen containing cisplatin (CDDP) or carboplatin and to define the safety profile of each arm of the above mentioned regimens in these patients

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years, with locally advanced, recurrent or metastatic endometrial adenocarcinoma, histologically diagnosed; at least 1 bidimensionally measurable lesion (> or =to 2 cm on computed tomography [CT]/magnetic resonance imaging [MRI] or > or =to 1 cm clinical lymph node confirmed by ultrasound or > or =to 1 cm skin lesion confirmed by photograph with ruler) located in a non-irradiated area measured less than 2 weeks before inclusion, according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC).
* Patients previously treated for locally advanced/metastatic disease with chemo-radiotherapy (total CDDP dose > or =to 100 mg/m2) or chemotherapy containing CDDP or carboplatin with at least 4 weeks' washout period from discontinuation of prior chemotherapy and fully recovered from toxic effects of prior chemotherapy (except for symptomatic peripheral neuropathy < or =to NCI-CTC grade 1 or alopecia).
* Patients with clinically or radiologically documented PD or recurrence during or after last chemotherapy and hormone therapy (hormone therapy stopped before study entry), Eastern Cooperative Oncology Group performance status (ECOG PS) < or =to 2, life expectancy > or =to 3 months, adequate bone marrow reserve, normal renal and liver function (neutrophil count > or =to 2000/mm³; platelet count > or =to 100 000/mm³; creatinine levels < or =to 1.5 x the upper limit of normal [ULN] of institutional values or creatinine clearance > 60 mL/min; total bilirubin level < 1.5 x ULN; [alanine amino transferase/aspartate amino-transferase < 2.5 x ULN without liver metastases, < 5 x ULN with liver metastases]).
* Laboratory values obtained in the week preceding study entry.
* Signed informed consent (prior to all study procedures)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-01; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Overall RR (World Health Organization [WHO]/Union Internationale Contre le Cancer [International Union Against Cancer] [UICC] criteria | during the study conduct

SECONDARY OUTCOMES:
Progression free-survival, duration of response and overall survival. | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Billon, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France